CLINICAL TRIAL: NCT05448690
Title: Comparative Effectiveness of Different Surgical Approaches for Giant Pituitary Adenomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Prof, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-060
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-combined approach (Single or Staged) (Active Comparator): Patients underwent transnasal approach or craniotomy approach; Patients underwent an initial surgery and a sencond staged surgery several months after the initial surgery
  Interventions: Procedure: Non-combined approach
- Combined approach (Experimental): Patients underwent a combined approach using transnasal approach and craniotomy approach simultaneously
  Interventions: Procedure: Two different approaches

INTERVENTIONS:
Procedure: Two different approaches — Please refer to Groups
  Arms: Combined approach
Procedure: Non-combined approach — Either transnasal, transcranial or a staged approach
  Arms: Non-combined approach (Single or Staged)

SUMMARY:
The surgical treatment strategy for giant invasive pituitary adenoma is one of the current hot spots in the field of clinical research on pituitary adenoma. A comprehensive literature search resulted in numerous previous studies to investigate the efficacy, advantages and disadvantages of different surgical options.

A single approach (transnasal or craniotomy) is theoretically less invasive and has a shorter hospital stay for the patient, but may result in postoperative bleeding due to residual tumor and damage to the intracranial vessels adhering to the tumor.

The advantage of the combined approach is that the tumor can be removed to the greatest extent possible. In addition, postoperative suprasellar hemorrhage can be prevented by careful hemostasis or intracranial drainage by the transcranial team if necessary. In this way, the risk of postoperative bleeding due to residual tumor can be significantly reduced.

In some cases, waiting a few months after the initial surgery for a second-stage procedure may also be an option when the patient's condition does not allow for a combined access procedure, when the tumor is hard, or when the blood preparation is insufficient. However, staged surgery increases the financial burden on the patient, and local scar formation may make second-stage surgery more difficult and decrease the likelihood of endocrine remission of functional pituitary tumors.

Given the complexity of the treatment of giant invasive pituitary adenoma, there is a need to conduct studies comparing the combined transnasal cranial approach, the single access transnasal or cranial approach, and the staged approach simultaneously to assess whether the combined transnasal cranial approach is superior to the single access transnasal or cranial approach or the staged approach in improving the tumor resection rate in giant invasive pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Giant pituitary adenoma (> 4cm in diameter)

Exclusion Criteria:

* most of the tumor were in the sellae, sphenoidal sinus or clivus.
* patients with craniopharyngioma or meningioma.

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Extend of resection | One month after surgery
  how much tumor was resected

SECONDARY OUTCOMES:
Risks | One month after surgery
  Proportion of Participants with hemorrage, infection or cranial nerve defect
Relapse or Mortality | From date of surgery until the date of first documented date of death from any cause, assessed up to 3 months after surgery
  Death from any cause
Karnofsky performance score | Three months after surgery
  Ranged from 0 to 100, the higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Chongqing People's Hospital, Chongqing, Chongqing Municipality
  - The first affliated hospital of Fujian Medical Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - General hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Renji Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - The first hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The first affliated hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qiao N, Gao W, Deng X, Xin T, Zhang G, Wu N, Wang P, Bi Y, Cong Z, Zhou Z, Li J, Sun S, Li M, Tang W, Yan X, Wang W, Qiu W, Yao S, Ye Z, Ma Z, Zhou X, Cao X, Shen M, Shou X, Zhang Z, Wu Z, Chu L, Qiu Y, Ma H, Wu A, Ma C, Lou M, Jiang C, Wang Y, Zhao Y. Combined simultaneous transsphenoidal and transcranial regimen improves surgical outcomes in complex giant pituitary adenomas: a longitudinal retrospective cohort study. Int J Surg. 2024 Jul 1;110(7):4043-4052. doi: 10.1097/JS9.0000000000001330. PMID 38498406